CLINICAL TRIAL: NCT03568396
Title: Validation of Pupillary Response to Nociceptive Stimulation in Cardiac Surgery During Extracorporeal Circulation Period
Acronym: DOLOCEC
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI18-DOLOCEC; 2018-A01137-48 (Other: IdRCB); 28/18_3 (Other: CPP)
Record Dates: First submitted 2018-06-08; First posted 2018-06-26 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Pupil; Analgesics; Opioid Use; Dose-Response Relationship, Drug; Anesthetics, Intravenous; Surgery, Cardiac; Circulation, Extracorporeal; Electric Stimulation; Electroencephalography/Drug Effects; Monitoring, Intraoperative; Adult; Remifentanil
Keywords: Nociceptive stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pupillometry: The relationship between the target effect site concentration of remifentanil and the pupil diameter and reactivity in response to a standard noxious stimulus.
  Interventions: Device: Pupillometer

INTERVENTIONS:
Device: Pupillometer — Measurement of pupil diameter and reactivity in response to a standard noxious stimulus in cardiac surgery during extracorporeal circulation period.

SUMMARY:
The relationship between the target effect site concentration of remifentanil and the pupil diameter and reactivity in response to a standard noxious stimulus in cardiac surgery during extra corporeal circulation will be evaluated.

DETAILED DESCRIPTION:
Anaesthesia will be induced with propofol to obtain loss of consciousness LOC in 30 patients who will undergo cardiac surgery requiring extracorporeal circulation and standardized support will be given to them till the extracorporeal circulation period. Thereafter, remifentanil will be titrated by increments of 0,5, from 1 up to 5 ng ml-1 during the extra corporeal circulation period. In the awake state, at LOC and at each plateau level of remifentanil CeT, mean arterial pressure, and BIS will be recorded. Pupil size and dilatation after a 60 mA, 100 Hz tetanic stimulation will be measured at LOC and at each plateau level of remifentanil.

ELIGIBILITY:
Inclusion Criteria:

* general anesthesia for cardiac surgery programmed requiring the realization of a sternotomy and the use of extra corporeal circulation
* age> 18 years

Exclusion Criteria:

* contraindication to the use of the products defined in the protocol of anesthesia (alprazolam, remifentanil, propofol, atracurium)
* sedation in progress with use of morphinomimetics
* urgent surgery
* preoperative existence of circulatory assistance
* preoperative existence of an intra-aortic balloon pump,
* bilateral ocular pathology (severe cataract, amblyopia, glaucoma, keratitis, conjunctivitis) and / or history of bilateral ocular surgery affecting the iris
* history of epilepsy, cerebral palsy
* peripheral neuromuscular diseases
* pathology with dysautonomia impairing the pupillary dilation reflex: insulin-dependent type 1 or type 2 diabetes with diabetic retinopathy, multiple sclerosis, systemic amyloidosis, uncontrolled hypertension, advanced Parkinson's disease
* ongoing treatment interfering with the autonomic and central nervous system likely to alter the pupillary dilation reflex: antiemetic (droperidol, metoclopramide), alpha-2 agonist (clonidine, dexmedetomidine), high doses of nitrous oxide
* treatment with severe anticholinergic effect: such as amitriptyline, amoxapine, atropine, benztropine, chlorpheniramine, chlorpromazine, clemastine, clomipramine, clozapine, darifenacin, desipramine, dicyclomine, diphenhydramine, doxepin, flavoxate, hydroxyzine, hyoscyamine, imipramine, meclizine, nortriptyline, orphenadrine, oxybutynin, paroxetine, perphenazine, procyclidine, promazine, promethazine, propentheline, pyrilamine, scopolamine, thioridazine, tolterodine, trifluoperazine, trihexyphenidyl, trimipramine
* pregnant or lactating women
* Patient having objected to the processing of his data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting for a general anesthesia for cardiac surgery programmed requiring the realization of a sternotomy and the use of extra corporeal circulation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Validation the use of pupillometry as a method of evaluation of nociception in cardiac surgery during the extracorporeal circulation period. | During surgery / one day
  To prove the existence of a linear correlation between the change in pupillary diameter and the concentration of remifentanil in cardiac surgery during the extracorporeal circulation period

SECONDARY OUTCOMES:
Validity of pupillometry nociception measurements in moderate hypothermia | During surgery / one day
  To prove existence of a linear correlation between the change in pupillary diameter and the remifentanil concentration in moderate hypothermia.

OTHER OUTCOMES:
Comparison of changes in mean arterial pressure and bispectral index to changes in pupillary diameter | During surgery / one day
  Compare changes in mean arterial pressure and bispectral index at the time of nociceptive stimulus with changes in pupillary diameter

CONTACTS AND LOCATIONS:
Overall Officials: Fabien ESPITALIER, M.D, Principal Investigator — University Hospital, Tours
Locations (1):
- Location Anesthesia-Resuscitation Department, University Hospital, Tours, Tours, France

IPD SHARING:
Plan to Share IPD: No